CLINICAL TRIAL: NCT01511861
Title: Assessing the Reliability of Non-invasive Blood Glucose Monitoring Device
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: GlucoVista (Industry)
Responsible Party: Sponsor
Other Study IDs: gluco02
Record Dates: First submitted 2012-01-13; First posted 2012-01-19 (Estimated); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Adequate glycemic control in patients with Diabetes Mellitus (DM) is a desired therapeutic goal that is difficult to achieve with current blood glucose monitoring technology. Home blood glucose monitoring (HBGM) technology, which requires finger pricking, is a source of severe inconvenience and hence, a lack of compliance.Thus, the need for non-invasive and easy to operate glucose monitoring in DM patients for strict glycemic control cannot be overemphasized.

The Glucometer GM-205 blood glucose readings are accurate and measure blood glucose with an acceptable mean relative error when compared to acceptable invasive blood glucose measurements.

The primary objectives of the trial are to determine:

1. Assessing the reliability of the Glucometer GM-205 in evaluating blood glucose levels compare to the standard glucose blood test
2. Creating database of glucose levels readings utilizing the Glucometer GM-205.

ELIGIBILITY:
Inclusion Criteria:

1. Diabetes Mellitus type one or type two.
2. Patients that are using Insulin.

Exclusion Criteria:

1. Vascular diseases
2. Pregnant and lactating women.
3. Exclusive use of long term Insulin.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with diabetes mellitus type 1 or type 2.
Sampling Method: Probability Sample
Enrollment: 137 (Estimated)
Dates: Start 2010-11; Primary Completion 2012-12 (Actual); Study Completion 2021-12 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Edith Wolfson Medical Center, Holon, Israel